CLINICAL TRIAL: NCT02058940
Title: Intravenous Exenatide Infusion in Critically Ill Patients With Acute Brain Injury
Brief Title: Intravenous Exenatide in Patients With Acute Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: AstraZeneca (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-1391; Astra Zeneca Pharmaceuticals (Other Grant/Funding Number: D5550L00025/ISSEXEN0038); Medtronic MiniMed, Inc (Other Grant/Funding Number: NERP14-008)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2017-09

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exenatide (Experimental)
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 50 ng/min IV for 30 minutes, then start 25 ng/min IV for a maximum duration of 48 hours

SUMMARY:
The purpose of this study is to assess the feasibility of exenatide infusion for the treatment of high blood sugars following acute brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Acute brain injury resulting in admission to the Neurosciences Intensive Care Unit for an anticipated length of stay >48 hours
* Two Blood glucose concentrations > 150 mg/dL and ≤300 mg/dL
* Informed consent obtained via proxy

Exclusion Criteria:

* Pregnant (verified by urine or serum pregnancy test within 24 hours of initiation of infusion) or lactating females
* Type 1 diabetes mellitus
* History of pancreatitis or risk factors for acute pancreatitis (i.e ethanol abuse, gall stones)
* Renal insufficiency defined as creatinine clearance (CrCL) < 45 mL/min
* Known history of gastroparesis
* History of surgery on stomach, esophagus or duodenum
* Diabetic Ketoacidosis or Hyperosmolar Hyperglycemic Nonketotic Syndrome
* Concurrent steroid use or planned post-operative steroid use
* History of organ transplantation
* Brain death or suspected imminent brain death within the next 72 hours
* Refractory intracranial hypertension defined as intracranial pressure (ICP) > 25 mmHg for greater than 15 minutes and refractory to medical intervention
* Currently enrolled in another investigational drug or device protocol
* Insulin infusion within 3 hours of study drug administration or confirmed long acting insulin or sulfonylurea use prior to admission within 24 hours of study drug administration
* Known allergy to exenatide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R. Pinelli, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina; UNC Medical Center, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exenatide
Started | 8
Completed | 7
Not Completed | 1
Not completed — Discharged from Critical Care Unit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exenatide
Number analyzed (Participants) | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.0 [58.8 to 67.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Primary Admitting Diagnosis [Count of Participants; unit: Participants]
  Intracerebral Hemorrhage | 3
  Acute Ischemic Stroke | 3
  Subarachnoid Hemorrhage | 1
  Subdural Hematoma | 1
Glasgow Coma Scale (GCS) [Median (Inter-Quartile Range); unit: units on a scale] — The Glasgow Coma Scale (GCS) aims to give a reliable and objective way of recording the conscious state of a person in response to defined stimuli. A patient is assessed against criteria of the scale, and the resulting points give a patient score between 3 and 15. Lower scores reflect a deeper state of unconsciousness.
  units on a scale | 10.5 [7.0 to 14.0]
Sequential Organ Failure Assessment (SOFA) [Median (Inter-Quartile Range); unit: units on a scale] — Sequential Organ Failure Assessment (SOFA) score evaluates six systems: respiratory, cardiovascular, coagulation, hepatic, renal and neurological. Each system gets a score from 0 (normal) to 4 (abnormal) and the sum of each score defines the final SOFA score, where 24 is the maximum score (high risk of mortality) and 0 is the minimum score (low risk of mortality).
  units on a scale | 2.0 [1.0 to 4.0]
Hunt and Hess Scale [Number; unit: units on a scale] — The Hunt and Hess scale is one of the grading systems used to classify the severity of a subarachnoid hemorrhage. It gives an index of the mortality associated with the various grades. The mortality is lowest with grade 1 and highest with grade 5. Population: Hunt and Hess Grade is only reported for patients with an admitting diagnosis of Subarachnoid Hemorrhage
  units on a scale
    number analyzed (Participants) | 1
    (all) | 2.0
Modified Fisher Grade [Number; unit: units on a scale] — The Modified Fisher Grade classifies the appearance of subarachnoid hemorrhage on CT scan. The appearance of the hemorrhage is determined on a scale of 0 (none evident) to 4 (most severe). Population: Modified Fisher Grade is only reported for patients with an admitting diagnosis of Subarachnoid Hemorrhage
  units on a scale
    number analyzed (Participants) | 1
    (all) | 3.0
Intracranial Pressure [Median (Inter-Quartile Range); unit: mmHg] — Intracranial pressure (ICP) is the pressure inside the skull and thus in the brain tissue and cerebrospinal fluid (CSF). ICP is measured in millimeters of mercury (mmHg) and, at rest, is normally 7-15 mmHg. Population: ICP is only reported in patients with Subarachnoid Hemorrhage. No patients with an admitting diagnosis of Subarachnoid Hemorrhage received ICP monitoring as part of standard of care and therefore data is not reported.
Cerebral Perfusion Pressure [Median (Inter-Quartile Range); unit: mmHg] — Cerebral perfusion pressure, or CPP, is the net pressure gradient causing cerebral blood flow to the brain (brain perfusion). It must be maintained within narrow limits because too little pressure could cause brain tissue to become ischemic (having inadequate blood flow), and too much could raise intracranial pressure (ICP). Population: CPP is only reported in patients with Subarachnoid Hemorrhage. No patients with an admitting diagnosis of Subarachnoid Hemorrhage received CPP monitoring as part of standard of care and therefore data is not reported.
Past Medical History [Count of Participants; unit: Participants]
  Diabetes | 4
  Hypertension | 6
  Hyperlipidemia | 4
  Cardiovascular Disease | 5
  Chronic Kidney Disease | 3
  Heart Failure | 1
Hemoglobin A1c (%) [Median (Inter-Quartile Range); unit: percent] | 6.5 [5.5 to 7.3]
Glucose [Median (Inter-Quartile Range); unit: mg/dL] | 191.0 [159.0 to 224.0]
Intensive Care Unit (ICU) Day of Study Drug Administration [Count of Participants; unit: Participants]
  Day 1 | 4
  Day 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Critically Ill Patients With Acute Brain Injury Achieving Pre-specified Feasibility Criteria
Description: Feasibility is defined as the percentage of patients 1) experiencing severe hypoglycemia (<40 mg/dL); 2) achieving glucose measurements within goal (110-180 mg/dL); and 3) experiencing nausea requiring discontinuation of exenatide therapy. The pre-specified criteria for determining feasibility includes the following: 1) at least 75% of patients achieving glucose measurements within goal (110-180 mg/dL) and 2) no more than 25% of patients experiencing severe hypoglycemia (<40 mg/dL) or nausea requiring exenatide discontinuation.
Time Frame: Over 48 hours from infusion initiation
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide
Number analyzed (Participants) | 8
percentage of patients
  Percentage Experiencing Severe Hypoglycemia | 0
  Percentage Achieving Glucose within Goal | 87.5
  Percentage with Nausea Requiring Discontinuation | 0

2. Secondary Outcome: Median Glucose Concentration During Exenatide Infusion
Description: Calculated from hourly blood glucose samples starting at infusion initiation over 48 hours
Time Frame: Over 48 hours from infusion initiation
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Exenatide
Number analyzed (Participants) | 8
mg/dL | 137.0 [118.0 to 164.3]

3. Secondary Outcome: Percentage of Glucose Measurements Within Goal Range
Description: Percentage of glucose measurements within goal range is calculated as the number of glucose measurements within goal range (110-180 mg/dL) for all patients/total number of glucose measurements collected for all patients.
Time Frame: Over 48 hours from infusion initiation
Measure: Number; unit: percentage of measurements
Arm/Group | Exenatide
Number analyzed (Participants) | 8
percentage of measurements | 69.6

4. Secondary Outcome: Median Time to Reach Glucose Measurements Within Goal Range (110-180 mg/dL)
Description: Calculated from hourly blood glucose samples starting at infusion initiation over 48 hours
Time Frame: Over 48 hours from infusion initiation
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Exenatide
Number analyzed (Participants) | 8
minutes | 200.0 [72.5 to 270.5]

5. Secondary Outcome: Glycemic Variability
Description: Glycemic variability is defined as the standard deviation of glucose calculated from hourly glucose measurements starting at infusion initiation over 48 hours
Time Frame: Over 48 hours from infusion initiation
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Exenatide
Number analyzed (Participants) | 8
mg/dL | 22.2 [15.0 to 36.3]

6. Secondary Outcome: Median Insulin Use
Description: Calculated from number of insulin units administered over 48 hours starting at infusion initiation
Time Frame: Over 48 hours from infusion initiation
Measure: Median (Inter-Quartile Range); unit: units/kg
Arm/Group | Exenatide
Number analyzed (Participants) | 8
units/kg | 0.03 [0.0 to 0.3]

7. Secondary Outcome: Percentage of Patients Requiring Rescue Insulin Infusion Protocol
Description: Defined as the percentage of patients requiring an insulin infusion to control glucose concentrations during exenatide treatment
Time Frame: Over 48 hours from infusion initiation
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide
Number analyzed (Participants) | 8
percentage of patients | 0

8. Secondary Outcome: Percentage of Hypoglycemic Episodes (<80 mg/dL)
Description: Percentage of hypoglycemic episodes is calculated as the total number of glucose measurements <80 mg/dL for all patients/total number of glucose measurements collected for all patients.
Time Frame: Over 48 hours from infusion initiation
Measure: Number; unit: percentage of measurements
Arm/Group | Exenatide
Number analyzed (Participants) | 8
percentage of measurements | 1.2

9. Secondary Outcome: Percentage of Patients With >1 Episode of Hypoglycemia (<80 mg/dL)
Description: Calculated from hourly blood glucose samples starting at infusion initiation over 48 hours
Time Frame: Over 48 hours from infusion initiation
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide
Number analyzed (Participants) | 8
percentage of patients | 12.5

10. Secondary Outcome: Percentage of Patients Experiencing Metabolic Crisis
Description: Metabolic crisis is defined as cerebral microdialysate glucose concentration <0.7 mmol/L in combination with lactate pyruvate ratio >40. Calculated from hourly microdialysis samples starting at infusion initiation over 48 hours
Time Frame: Over 48 hours from infusion initiation
Population: No patients received invasive intracranial multimodal monitoring as a part of their standard of care, as such, these endpoints were not collected.
Arm/Group | Exenatide
Number analyzed (Participants) | 0

11. Secondary Outcome: Median Daily Intracranial Pressure
Description: Calculated from hourly measurements starting at infusion initiation over 48 hours
Time Frame: Over 48 hours from infusion initiation
Population: No patients with an admitting diagnosis of Subarachnoid Hemorrhage received ICP or CPP monitoring as part of standard of care and therefore data is not reported.
Arm/Group | Exenatide
Number analyzed (Participants) | 0

12. Secondary Outcome: Median Daily Cerebral Perfusion Pressure
Description: Calculated from hourly measurements starting at infusion initiation over 48 hours
Time Frame: Over 48 hours from infusion initiation
Population: as for outcome 11
Arm/Group | Exenatide
Number analyzed (Participants) | 0

13. Secondary Outcome: Percentage of Hypotensive Episodes (SBP<100 mmHg)
Description: Defined as the number of hypotensive episodes (SBP<100 mmHg)for all patients/total number of blood pressure measurements collected for all patients.
Time Frame: Over 48 hours from infusion initiation
Measure: Number; unit: percentage of measurements
Arm/Group | Exenatide
Number analyzed (Participants) | 8
percentage of measurements | 1.2

14. Secondary Outcome: Percentage of Patients With >1 Episode of Hypotensive Episode (SBP<100 mmHg)
Description: Calculated from blood pressure measurements starting at infusion initiation over 48 hours
Time Frame: Over 48 hours from infusion initiation
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide
Number analyzed (Participants) | 8
percentage of patients | 12.5

15. Secondary Outcome: Correlation of Exenatide Concentrations With Creatinine Clearance
Description: Spearman's correlation coefficient calculated from exenatide concentrations and urine creatinine measurements collected for all patients during the study period. A correlation coefficient is a numerical measure of some type of correlation, meaning a statistical relationship between two variables. Spearman's correlation coefficient assumes values in the range from -1 to +1, where +1 indicates the strongest possible agreement and -1 the strongest possible disagreement.
Time Frame: Over 48 hours from infusion initiation
Measure: Number; unit: correlation coefficient
Arm/Group | Exenatide
Number analyzed (Participants) | 7
correlation coefficient | -0.2
Statistical Analysis 1: Comparison: Exenatide; Test type: Other; p = 0.2, Spearman's Correlation Coefficient

16. Secondary Outcome: Exenatide Elimination Rate Constant After Discontinuation of Infusion
Time Frame: 24 hours
Population: The institutional review board requested the study team limit exenatide concentration sampling to during the infusion. Samples were not collected after discontinuation of study drug. As such, this pharmacokinetic parameter is not reported.
Arm/Group | Exenatide
Number analyzed (Participants) | 0

17. Secondary Outcome: Exenatide Area Under the Concentration-time Curve After Discontinuation of Infusion
Time Frame: 24 hours
Population: as for outcome 16
Arm/Group | Exenatide
Number analyzed (Participants) | 0

18. Secondary Outcome: Median Intensive Care Unit Length of Stay
Description: Defined as the number of days admitted to the Intensive Care Unit
Time Frame: From enrollment to 30 days post study drug discontinuation
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Exenatide
Number analyzed (Participants) | 8
days | 9.0 [7.8 to 14.8]

19. Secondary Outcome: Median Hospital Length of Stay
Description: Defined as the number of days admitted to the hospital
Time Frame: From enrollment to 30 days post study drug discontinuation
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Exenatide
Number analyzed (Participants) | 8
days | 12.5 [9.0 to 27.3]

ADVERSE EVENTS:
Time Frame: From study enrollment to 30 days post discontinuation of Exenatide, up to 1 month
Arm/Group | Exenatide
All-Cause Mortality (participants affected / at risk) | 3/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=8)
Death (Nervous system disorders) | 3 — All 3 patients completed study treatment. Cause of death due to underlying neurological injury with family deciding to place patients on comfort care.

LIMITATIONS AND CAVEATS:
Trial ended early and did not achieve targeted recruitment goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT02058940/Prot_SAP_000.pdf